CLINICAL TRIAL: NCT03049007
Title: The Aarhus Bereavement Study - a Prospective Study on Natural and Prolonged Grief Reactions in the Adult Population
Brief Title: The Aarhus Bereavement Study
Acronym: TABS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: AU2017
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Grief
Keywords: bereavement; natural grief; prolonged grief; complicated grief
MeSH Terms: interventions — Fertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Partner: Spousal bereaved individuals (age 25-85) in the Central Denmark Region identified through a data extraction of the Danish Civil Registration System (CPR) every sixth week over a period of one year. The group will complete a survey at respectively 2 (T1), 6 (T2), 11 (T3), 18 (T4), and 26 (T5) months post-loss as well as 3, 4, 5 and 6 years post loss.
  Interventions: Diagnostic Test: Survey
- Child: Parental bereaved individuals (age 18 or above) that are children of the partner group. The group will complete a survey at respectively 2 (T1), 6 (T2), 11 (T3), 18 (T4), and 26 (T5) as well as 3, 4, 5 and 6 years post loss.
  Interventions: Diagnostic Test: Survey

INTERVENTIONS:
Diagnostic Test: Survey — Completion of surveys with diagnostic measurements (e.g., PGD, depression, anxiety, PTSD).

SUMMARY:
Psychological distress is a natural reaction following the death of a loved one. Nevertheless, research has shown that for a significant minority of bereaved individuals the grieving process is disturbed. These individuals experience an intense grief reaction that persists across time characterized by longing for the deceased or persistent preoccupation with the deceased. It has been suggested that this intense, persistent grief reaction meets criteria to be considered a distinct mental disorder. Prolonged grief disorder (PGD) has been proposed to capture this condition and will be included in the forthcoming ICD-11. The proposed project aims to prepare healthcare services to use the diagnosis of prolonged grief disorder (PGD) by determining the frequency of PDG in a population sample of bereaved spouses and their adult children. It will also identify early predictors of PGD and trajectories of natural and prolonged grief as well as investigate the specificity of PGD in relation to other common loss-related reactions. Thus, the project will provide a prognostic tool to identify individuals with high versus low risk of developing PGD.

DETAILED DESCRIPTION:
BACKGROUND:

Prolonged grief disorder (PGD) is a new diagnosis that may occur after the death of a partner, parent, child, or other person close to the bereaved. PGD is characterized by a persistent and pervasive grief response including longing for the deceased or persistent preoccupation with the deceased accompanied by intense emotional pain (e.g. sadness, guilt, anger, denial, blame, difficulty accepting the death). The disorder has been admitted as an official diagnosis in the World Heath Organization's newest diagnostic manual (International Classification of Diseases, 11th revision; ICD-11). When introducing the diagnosis in ICD-11, health care services are obliged to identify and treat PGD.

PURPOSE AND AIMS:

The primary purpose of the study is to prepare healthcare services to use the diagnosis of PGD. More specifically, the project aims to determine the frequency and structure of PDG in a population sample of bereaved spouses and their adult children. It will also identify early predictors of PGD and common trajectories of natural and prolonged grief as well as investigate the specificity of PGD in relation to other common loss-related reactions. Finally, the project will also assess the socioeconomic costs of PGD by analyzing health data registries.

HYPOTHESES:

Based on existing bereavement literature and empirical research, the project explores the following hypotheses:

1. High rumination, low levels of mental and physical health, loss of spouse versus loss of parent, and presence of psychopathology at time of loss (T1) will predict degree of PGD symptoms among the bereaved at 6 (T2) and 11 (T3) months post-loss.
2. The majority of bereaved individuals will exhibit a grief trajectory with a gradual decline in PGD symptoms over time, while a significant minority of bereaved individuals will show a trajectory with high levels of PGD symptoms across all measured time-points.
3. PGD, PTSD, depression, and anxiety will be distinct constructs.

On a more genereal level. trajectories of grief and in line with the aim of this study, structure and frequency of prolonged grief disorder, and the relationship with PGD and other forms of complicated grief reactions will be analyzed across the timepoints and factors related to grief will be investigated.

PARTICIPANTS AND PROCEDURES:

Individuals (age 25-85) will be consecutively recruited through the Danish Civil Personal Registry (CPR) from the Central Region of Denmark. After the loss, participants are contacted with a letter of condolence and a brief introduction to the study. Two months post-loss, potential participants are telephoned and invited to participate in the study. Participants are asked to complete self-report questionnaires, respectively at 2 (T1), 6 (T2), 11 (T3), 18 (T4), 26 (T5), months and continue with data collections at 3 (T6), 4 (T7), 5 (T8) and 6 (T9) years post-loss. To meet different needs, participants can choose to fill in the questionnaire online or by postal service.

Bereaved individuals constitute a highly vulnerable group with a heightened risk of suicide, social isolation, depression, etc. In the event, participants appear suicidal or particularly distressed (e.g. high score on suicidal ideation) they will be contacted by the researchers and a suicide risk screening is performed.

ELIGIBILITY:
Inclusion Criteria, partner:

* Resident in the following municipalities: Aarhus, Favrskov, Horsens, Norddjurs, Odder, Randers, Silkeborg, Skanderborg, Syddjurs
* Age 25-85
* Has lost a partner or spouse within the last 5 weeks from inclusion

Inclusion Criteria, child:

* Resident in the following municipalities: Aarhus, Favrskov, Horsens, Norddjurs, Odder, Randers, Silkeborg, Skanderborg, Syddjurs
* Age 18-85
* Has lost a parent or step-parent within the last 5 weeks from inclusion

Exclusion Criteria, all:

- Psychiatric inpatients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Spousal bereaved individuals (age 25-85) living in the Central Denmark Region plus their adult children (age 18 or above). Eligible participants will be identified through a data extraction of the Danish Civil Registration System (CPR) every sixth week over a period of one year.
Sampling Method: Probability Sample
Enrollment: 1243 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Prolonged grief | 2, 6, 11, 18, and 26 months post-loss
  Changes in prolonged grief symptoms measured using the Prolonged Grief Disorder-13 (PG-13; Prigerson et al., 2009)
Complicated grief | 2, 6, 11, 18, and 26 months post-loss
  Changes in complicated grief symptoms measured using the Inventory of Complicated Grief Revised (ICG-R; Prigerson & Jacobs, 2001)

SECONDARY OUTCOMES:
Depression | 2, 6, 11, 18, and 26 months post-loss
  Symptoms of depression are measured using the Center for Epidemiologic Studies Short Depression Scale (CES-D 10; Radloff, 1977)
Generalized anxiety | 2, 6, 11, 18, and 26 months post-loss
  Symptoms of generalized anxiety are measured using the Generalized Anxiety Disorder-7 (GAD-7; Spitzer et al., 2006)
Post-traumatic stress | 2, 6, 11, 18, and 26 months post-loss
  Symptoms of post-traumatic stress are measured using the PTSD checklist - Civilian Version (PCL-C; Ruggiero et al., 1999)
Well-being | 2, 6, 11, 18, and 26 months post-loss
  Levels of well-being are measured using the World Health Organization-5 (WHO-5; Heun et al., 2001)
Mental and physical health | 2, 18, and 26 months post-loss
  Levels of mental and physical health are measured using the 12-Item Short Form Health Survey (SF-12; Ware et al., 1996)

OTHER OUTCOMES:
Loneliness | 2, 6, 11, 18, and 26 months post-loss
  Levels of loneliness are measured using the Three-Item Loneliness Scale (T-ILS; Hughes, Waite, Hawkley, & Cacioppo, 2004)
Rumination | 2, 6, and 11 months post-loss
  Levels of rumination are measured using the Rumination-Reflection Questionnaire (RRQ; Trapnell & Campbell, 1999)
Social support | 2, 6, and 11 months post-loss
  Levels of social support are measured using the Crisis Social Support scale (CSS; Joseph, Andrews, Williams, & Yule, 1992)
Attachment | 2 months post-loss
  Attachment orientations are measured using the Experiences in Close Relationship Scale - short (ECR; Wei et al., 2007)
Optimism | 2 months post-loss
  Levels of optimism are measured using the Life Orientation Test - Revised (LOT-R; Scheier, Carver, & Bridges, 1994)
Neuroticism | 2 months post-loss
  Levels of neuroticism are measured using the NEO Personality Inventory-Revised - neuroticism only (NEO-PI-R; Costa & McRae, 2004)
Centrality of event | 2, 6, and 11 months post-loss
  Levels of centrality of event are measured using the Centrality of Event Scale (CES; Berntsen & Rubin, 2006)
Emotional expression | 2 months post-loss
  Ability of emotional expression are measured using the Flexible Regulation of Emotional Expression (FREE; Burton & Bonanno, 2015)
Emotion regulation | 2 months post-loss
  Levels of emotion regulation are measured using the Emotion Regulation Questionnaire (ERQ; Gross & John, 2003)

CONTACTS AND LOCATIONS:
Overall Officials: Maja O'Connor, MSc PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Department of Psychology and Behavioural Sciences, Unit for Bereavement Research, Aarhus, Denmark

REFERENCES:
- [Derived] Komischke-Konnerup KB, Vang ML, Lundorff M, Elklit A, O'Connor M. Do early symptoms of prolonged grief disorder lead to symptoms of posttraumatic stress disorder and depression? A longitudinal register-based study of the two first years of bereavement. J Psychopathol Clin Sci. 2023 Nov;132(8):996-1006. doi: 10.1037/abn0000859. Epub 2023 Aug 3. PMID 37535580
- See also: Webpage with information on the research unit conduction the study — https://psy.au.dk/en/research/research-centres-and-units/unit-for-bereavement-research